CLINICAL TRIAL: NCT02118454
Title: ART Adherence Behaviour and Practices Among HIV Positives in Kolkata, India-a Pilot Project
Brief Title: Antiretroviral Adherence and Quality-of-life Support for HIV+ Patients in India With Twice-daily Interactive Voice Response (IVR) Calls With Health and Mental Health Messaging Compared to Weekly IVR Survey Only Control Condition: The Mobile-messaging Adherence and Support for Health Study, India.
Acronym: MASHIndia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Indian Council of Medical Research (Other Government); Durbar Mahila Samanwaya Committee (Unknown); Calcutta School of Tropical Medicine (Other); Dimagi Inc. (Industry)
Responsible Party: Principal Investigator, Dallas Swendeman, Assistant Professor-in-Residence, Center Co-Director, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R21AI094666 (NIH); INDO-US/86/9/20 1O-ECD-II (Other Grant/Funding Number: Indian Council of Medical Research [ICMR] Grant Number)
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: HIV/AIDS
Keywords: Medication adherence; Self-management; Depression; Coping; Social support; Mobile health; Antiretroviral treatment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily IVR calls (Experimental): The Daily IVR Calls Intervention: consisting of two (2) automated voice calls ("intervention messages") each day for six months, PLUS one IVR assessment call (consisting of four [4] questions) every week for 6 months
  Interventions: Behavioral: Daily IVR Calls Intervention
- Weekly IVR Survey Only (Active Comparator): The Weekly IVR Survey Only control condition: consisting of standard care, PLUS one IVR assessment call (consisting of four [4] questions) every week for 6 months.
  Interventions: Behavioral: Weekly IVR Survey Only

INTERVENTIONS:
Behavioral: Daily IVR Calls Intervention
  Arms: Daily IVR calls
Behavioral: Weekly IVR Survey Only
  Arms: Weekly IVR Survey Only

SUMMARY:
The purpose of this study is to test whether twice-daily Interactive Voice Response (IVR) calls made at the estimated times of patients' antiretroviral (ART) medication dosing and three reminder calls for monthly clinic appointments, will result in improvements in ART adherence, appointment attendance, health indicators (CD4 cell counts), coping skills, social support, depressive symptoms, and other quality-of-life indicators, compared to a control group receiving one IVR assessment call each week, over six months.

This is a randomized controlled trial of the IVR intervention with n=400 PLH taking first line ART in India on a twice-a-day dosing schedule. The research is supported by an Indo-U.S. Bilateral review and funding collaboration between NIH and ICMR. The research is being implemented in Kolkata by Drs. Smarajit Jana (PI, India) and Protim Ray (Project Director) at Durbar, a community-based organization providing HIV/STD prevention and community development programs with sex workers and other at-risk communities.

This is Phase 2 of a two-phase pilot project. Phase 1 was a one-month no-control pilot (n=46) for feasibility, acceptability, and patient feedback on preferences for messaging content. Phase 2 has two sites, described as Phases 2A and 2b, which will occur simultaneously and differ only in their recruitment sites and corresponding sampling strategy (sample size, gender ratio, eligibility criteria) based on site population characteristics.

* Phase 2A will recruit n=80 women and n=20 men from Durbar's Mamata Care and Treatment Center (MCTC) (providing HIV testing and treatment linkage and support) and associated Mamata Network of Positive Women (MNPW), which focus on HIV+ sex workers and their male partners and networks.
* Phase 2B will recruit n=100 women and n=200 men from the ART Centre at the Calcutta School of Tropical Medicine (STM), which hosts the largest ART center in the Northeast Region of India and has over 3,000 active patients on first line ART.

The sampling plan reflects the gender distribution of clients and patients at the two sites.

Participants will be randomized within each site and gender sub-sample to receive:

* The IVR Intervention: consisting of two (2) automated voice calls ("intervention messages") each day for six months, PLUS one IVR assessment call (consisting of four [4] questions) every week for 6 months; OR,
* The Control Condition: consisting of standard care, PLUS one IVR assessment call (consisting of four [4] questions) every week for 6 months.

All participants will be interviewed in-person by a research team member at baseline and followed-up at 2- 4- and 6-months using structured questionnaires and recording information from the participant's personal medical record (i.e., their "ART Card") to assess background characteristics and intervention impacts on ART adherence, health quality-of-life (i.e., depressive symptoms, social support). All participants will receive one IVR assessment phone call (consisting of four (4) questions during each week of the 6 month study. Each once-a-week IVR assessment will ask about missed medication and the participant's health/quality of life, and participants will respond by keying in a 1 (yes) or 2 (no) on their mobile phone.

DETAILED DESCRIPTION:
The originally proposed study aims were revised slightly during the review process from the Indian Council of Medical Research (ICMR), which is NIH equivalent and partner funder of this research (see "ICMR Comments" document). The original proposal examined comprehensive messaging for adherence, risk reduction, and quality of life (i.e., emotional support), compared to medication adherence messages only. The protocol was revised to compare comprehensive messaging to standard care. The IVR intervention is built on Dimagi's original ART adherence text-messaging support system called "ARemind". Therefore, the aims of this study are to:

1. Adapt the ARemind mobile phone ART adherence mobile phone messaging system for PLH in Kolkata, India;
2. Further develop ARemind to address the co-occurring factors of ART non-adherence, poor mental health, and transmission risks;
3. Examine the acceptability, engagement, and adherence by PLH to the IVR messaging system; and
4. Examine the efficacy of the twice daily ART reminder calls with health messages compared to standard care, for medication adherence only compared to standard care to improve adherence and mental health, and reduce transmission risks, in a randomized controlled trial.

BACKGROUND The 2.3 million persons living with HIV (PLH) in India are being offered access to anti-retroviral therapies (ART) by the government. ART offers the possibility of improving health and reducing HIV transmission by decreasing HIV viral loads in PLH. Yet, non-adherence remains high globally, with an estimated 50% of PLH in India not maintaining adherence to 95% of ART doses, which is considered the adherence rate needed to maintain HIV viral suppression.

Mobile phones have been used in the US and globally to increase ART adherence among PLH. As a low cost, easily diffused intervention strategy in a country such as India in which the mobile phone penetration rate is expected to reach 100% by 2014 (Informa World, 2010), designing a mobile phone intervention to increase ART adherence is a potentially highly efficacious intervention.

However, because HIV is a chronic infectious disease, PLH are also challenged with maintaining mental health and reducing transmission risks (Swendeman et al., 2009a). Furthermore, reviews and meta-analyses have concluded that ART adherence interventions are more effective when a comprehensive approach is adopted (Malta, 2008; Rueda, 2006; Simoni, 2006). In particular, mental health symptoms and transmission acts that co-occur with and undermine ART adherence (Kalichman, 2008, Malta, 2008) are likely to be behaviors that may also be influenced by mobile phone delivered interventions. Thus, this study aims to adapt and develop an intervention to improve and maintain medication and appointment adherence, reduce transmission acts, and improve quality of life including mental health symptoms.

Phase 1 pilot testing (June - August, 2013) was recently completed by the research team in Kolkata with PLH (n=46) taking ART and clients of Durbar's Mamata Care and Treatment Center (MCTC), members of Durbar's "Mamata Network of Positive Women" (MNPW), and their peers. Phase 1 involved a 1-month pilot test of the IVR messaging intervention, including baseline and a follow up assessment, and brief open-ended feedback interview and focus group feedback interviews at the follow up to inform the current protocol.

Three world-renowned HIV prevention and technology organizations will collaborate in Phase 2 research activities: 1) UCLA Center for HIV Identification, Prevention, and Treatment Services (CHIPTS), with expertise in behavioral intervention development, adaptation, and randomized trials for PLH and other high-risk populations; 2) Durbar, with expertise in multi-level prevention and support services for high-risk populations in India; and 3) Dimagi Inc., a technology company with expertise in mobile phone solutions for global health challenges. Dimagi developed "ARemind" to assess and remind ART and appointment adherence with feedback from PLH and providers in the U.S. and tested in a pilot study and prior NIH-funded grants. The software reminds PLH through text-messaging (i.e. Simple Messaging Service [SMS]) or Interactive Voice Response (IVR) methods. This program can also be leveraged to address the co-morbid challenges of preventing transmission and improving mental health and quality of life for PLH. In this study, ARemind will be adapted and developed for PLH recruited from two sites in Kolkata, India; 1) a community based care and treatment center operated by Durbar serving primarily female sex workers living with HIV (i.e., the Mamata Care & Treatment Center [MCTC] & Mamata Network of Positive Women [MNPW]), and 2) PLH recruited from the primary ART Centre at the Calcutta School of Tropical Medicine (STM).

DESIGN AND METHODS After recruitment and consenting into Phase 2, participants will be randomized within site and gender sub-samples to either intervention or standard care (control) conditions and complete the Phase 2 Baseline Survey. Participants who do not have their own personal mobile phone will be provided with a mobile phone and phone line (i.e., Sim card) with service paid for by the research team during the 6-month study period. All participants will complete in-person follow up interviews (with a research team member) every two months for six months, which include medical record abstraction, and brief weekly IVR assessments (on their own, via their mobile phone). Study documents and IVR messages will be available in Bengali and Hindi.

RECRUITMENT The source of referrals will be MCTC staff or clients or MNPW network members or their peers (Phase 2A), or STM ART Centre staff, patients or their peers (Phase 2B). Staff, patients, or clients at from any of these sites will have recruitment scripts administered to them by a member of the research team and will be provided with study information cards to give to their patients, clients, or peers who they think may be interested in participating in the research study. If the patient, client or peer is interested in finding out more about the study, they will contact the research team directly using the phone number on the study information cards.

A member of the Durbar MCTC Staff (Phase 2A) or STM Staff (Phase 2B) will administer a verbal introduction script to patients in the waiting areas of the MCTC or STM. MCTC client flow is modest, seeing less than a dozen PLH each day. STM patient flow sees hundreds of 1st-line ART patients each day, with long lines and waiting times to see the physicians, lab technicians, counselors, and to receive ART refills. The introduction script tells the patients/clients where the recruiters are from and that they are part of a research study. Next a research team member will describe the study to the people sitting in the waiting areas. If a potential participant is interested in hearing more from the team member, they will go to a private office within the MCTC (Durbar office - Phase 2A) or STM (Study office provided by the STM - Phase 2B) where the research team member will administer the screening questions.

SCREENING [In-Person] If the patient, client, or peer is interested to find out if s/he is eligible to participate based on the (introductory) recruitment script, the research team member will privately administer the screening questions. If eligible based on self-report, eligibility will be confirmed by the study staff reviewing the potential participant's ART Card. Responses will be recorded in the Dimagi phone application by the study staff.

[By Telephone] If the caller is interested to find out if s/he is eligible to participate based on the (introductory) recruitment script, the research team member will administer the screening questions. If the potential participant is eligible based on their self-report, an in-person meeting will be scheduled at the MCTC or STM study offices. The screening questions will be re-administered at the in-person meeting, confirmed by review of the ART Card, and responses recorded in the Dimagi phone application by the study staff.

Durbar Staff will screen potential participants in a private room or private area at the School of Tropical Medicine or the MCTC at Durbar. Self-report by potential participants of the following information will determine their preliminary eligibility: 1) Age; 2) how long on ART; 3) which ART regimen (1st, 2nd, 3rd line); 4) if received CD4 count result in past two months (for Phase 2A at MCTC/MNPW) or past 2 months (for Phase 2B at STM); and 4) if missed taking any ART doses in the past 6 months. If eligible based on self-report, verbal consent will be obtained to review the potential participant's ART Card to confirm eligibility by checking: 1) identity from photo, 2) Age, 3) how long on ART, 4) which ART regimen (1st, 2nd), and 5) date of last CD4 count result. All screening information except for identity (photo, name) but also including gender, language, and literacy (literate or not) will be recorded on the Screening Questionnaire in order to compare ineligibles, those who do not consent to participate, and consented participants. Screening data are entered into a secure database in the Dimagi system using the study staff mobile phones with the Dimagi application.

CONSENT & ENROLLMENT If recruitment/screening is in-person, eligible participants will be asked if they want to enroll in the study at that time. If they do, the research team member will administer the Informed Consent Form. If recruitment/screening in over the telephone, the research team member will make an in-person appointment with the eligible participant to repeat the screening, confirm eligibility based on ART Card review, and administer the Informed Consent Form, if the eligible participant wants to enroll in the study.

BASELINE AND FOLLOW UP SURVEY INTERVIEWS Study interviewers will use mobile phones with a survey application programmed by Dimagi to administer the baseline and follow-up surveys to participants and record their responses. The Baseline and Follow-Up interviews at 2-, 4-, and 6-months will generally be scheduled on the same day as a medical visit at STM ART Centre, or shortly after an ART Centre visit if the participant was recruited from MCTC/MNPW.

ART MEDICAL CARD ABSTRACTION All ART patients in India keep their own medical record and carry it with them to their monthly appointments for check-ups and medication refill. The "ART Card" includes the patient's name, photo, date of birth, address, phone numbers, contact names and phone numbers, and information related to HIV treatment outcomes, including CD4 cell counts (conducted once every 6 months) and ART pill counts (i.e., an estimate of adherence) collected at each monthly clinic visit. (The STM ART clinic also keeps a copy of the record). During Screening and Baseline and Follow-Up surveys the ART Card will be reviewed by the study interviewer to confirm the participant's identity and eligibility, and then to record the participant's CD4 and ART pill counts and their dates in the survey application. At Baseline, the prior two CD4 and prior 6 ART pill counts will be recorded. At follow-up interviews the prior two pill counts and any new CD4 count will be recorded.

WEEKLY IVR ASSESSMENT CALLS All participants will receive one IVR Assessment call each week that consists of four questions, one on medication adherence, two on depressive symptoms, one on physical symptoms. Responses are entered by pressing 1 (yes) or 2 (no) on the phone keypad. Once a response is received, the next question plays. If an IVR assessment call is not answered, the system attempts 3 repeat calls within one hour of the specified call time. If participants do not respond to 2 consecutive weeks' IVR assessment calls, a study interviewer will call the participant's phone (and other contacts, if needed) to confirm that the mobile phone service is still active and remind the participant how the IVR system functions.

Participants select the day and time to receive the IVR assessment calls, which they confirm or change at each follow up interview or can change by calling the study contact number. If participants request it, they can decline to receive IVR assessment calls. Female participants will receive calls with a female voice and vice versa for male participants.

Feedback from the PLH CAB, service providers, another similar study in India, and our Phase 1 experience found that reading and technological literacy are low enough among some PLH that this interactive feature may prove unreliable. Therefore, participants will receive a brief training from the study interviewer at the baseline meeting on how the IVR assessment calls function and how to respond using the keypad.

INTERVENTION: IVR MESSAGING SYSTEM The IVR messaging system automatically sends pre-recorded voice messages twice each day, once in the morning and once in the evening, to participants in the intervention condition. The call times are linked to the times that a participant reports typically taking his/her ART medication (twice a day is the standard dosing schedule for 1st-line ART) or at an alternative time that the participant specifies in the Baseline and Follow-Up Surveys. The most basic function of the calls is to act as "alarm reminders" to take ART, whether or not a call is answered, while the messaging content has a dual function of being engaging for participants and potentially impacting other study outcomes beyond ART adherence. Messaging automatically stops after the 6-month follow up is completed or when a participant declines receiving messages or withdraws from the study.

The IVR intervention messages are less than 60 seconds each and focus on several key domains identified is being important and engaging by the target population and by the intervention team: 1) Illness-related information (i.e., TB, malaria, but no HIV-specific messages) and self-management strategies for medication adherence and symptom/side-effect management (nausea, diarrhea, dehydration); 2) Wellness-related messages focused primarily on diet, nutrition, and hygiene; and 3) Mental health related messages focused on self-management strategies for stress-reduction, mood improvement, positive cognitions, and social support. Not all message content is being evaluated by corresponding outcome measures. Specifically, change in knowledge is not being assessed in order to reduce assessment burden and focus on behavioral outcomes. The functional role of some messages is intended for engagement, intervention framing, and motivation, in addition to behavioral cues. Over 120 messages were developed, split about evenly across the three categories of illness, health, and mental health messages. Messages were randomly sorted within each category and then sequenced in an alternating order for the final message delivery queue. The number of messages was selected to not have any message repeat over two months.

HIV & STI "Specific" Messages Phase 1 results identified that some PLH preferred specific messages about HIV/AIDS and risk behaviors, while others, particularly those with children, preferred only general health messages to protect their privacy in the event someone else answered the phone call. Therefore, from Baseline to the 2-month follow-up assessment, participants will not receive messages that specifically mention HIV/AIDS or sexual behaviors or sexually transmitted infections (STI), which we refer to as "Specific" messages. Specific messages are intentionally not implemented from Baseline to 2-month follow up to allow participants to actually experience the intervention modality before opting to receive specific messages that might result in adverse events such as HIV disclosures. At 2-month and 4-month follow-up interviews participants can "opt-in" to receive "Specific" messages for the following two months, with messaging preferences recorded in the survey application and automatically linked to the Dimagi messaging system. Specific message libraries are currently being prepared. Participants in the Intervention Condition will be able to opt-out of receiving specific (i.e. HIV-related) IVR messages at any time by calling the study team.

ART Clinic Appointment Reminders The IVR messaging system also sends ART clinic appointment reminders for the ART Centre visit scheduled for 8-weeks (2-months) after the baseline, 2-month, and 4-month follow-up interviews, or at a more specific date provided by the participant. ART Centre follow-up visits are typically scheduled exactly four weeks apart. The appointment reminder will be sent in the morning call 7 days in advance of the appointment and again 2 days in advance. If the appointment reminder calls are not answered, the system attempts 3 repeat calls within one hour of the specified call time and repeats at the subsequent specified call times until answered or until the day of the scheduled appointment.

"National Do Not Call" (NDNC) Registry: India has a "National Do Not Call" (NDNC) registry for cell phone numbers that is an "opt-in" registry. In order to be put on the NDNC registry, cell phone owners must contact the registry to have their cell phone number added. Once added, being on the NDNC registry prevents the cell phone from receiving "robo-calls" - typically commercial solicitations. Since this study's "IVR Messaging System" and "Weekly Assessment Calls" are technically "robo-calls," the participant (if using their own cell phone) must not be registered with the NDNC registry in order to participate in the study. If the participant has previously registered with the NDNC registry, we will get permission from the participant and assi ist them to remove their cell phone number from the NDNC registry for the duration of the study. At the study completion, if requested, the researcher will assist the participant to opt-in to the NDNC registry.

Message Monitoring and Follow Up The IVR system also monitors and reports through the Dimagi system to the study team whether each call was answered and the duration of the call to estimate whether it was listened to completely or not. Message monitoring reports will be generated on a weekly basis. If the reports indicate that calls are not being answered by a participant for two consecutive weeks at the phone number they specified, a study team member will call the participant's phone (and other contacts, if needed) to confirm service is still active or obtain a new preferred phone number from the participant (see Phone Follow-Up Script).

TIME FOR ASSESSMENT AND INTERVENTION ACTIVITIES Total study time is 6.5 hours for control group and 12.5 hours for the intervention group. The Baseline Interview, including informed consent and instructions, will last about 2 hours. The three Follow-up Interviews will last about 1 hour each. IVR Assessment messaging requires about 3 minutes for the participant to listen and respond to the messages each week for 6 months (about 1.5 hours). Intervention messaging requires about 2 minutes per day for x 6 months (about 6 hours).

DATA MANAGEMENT All data will be coded with a unique participant identification number (PID) generated by a computerized algorithm from the participant's name, father's name, age, sex, and phone numbers collected in the "Registration Information" section of the baseline interview. The interviews are conducted with computerized assessments using mobile phones programmed by Dimagi Inc., with data stored on their HIPAA compliant servers in the United States. The "Registration Information," which includes locator information (i.e., phone number and an alternate contact and phone number), will be stored in separate files from the interview data on the Dimagi servers, with different password-protected access controls and will only be accessible by the PI & other research team members. The "Registration Information" questions are repeated in the follow up interview to verify the participant's identity as a study participant. Only study staff will have access to the "Registration Information" via their study specific mobile phone and its installed assessment application from Dimagi, with the phone password protected and the Dimagi application also having a login ID and password.

Signed consent forms will be stored in a locked file in a locked office at the Durbar research office. All forms that record data in this study will be electronic and managed by Dimagi: 1) Screener data, 2) Locator Form (i.e. "Registration Form"), 3) Baseline and Follow-up survey data, and 4) IVR assessment data. At the completion of the study, all data will be downloaded by the UCLA research team and permanently deleted from the Dimagi servers.

DATA ANALYSES Baseline descriptive analyses will be conducted with simple frequency distribution methods (means, mode, ranges, standard deviations). Follow-up data will be examined with linear and logistic regression. Unadjusted and adjusted longitudinal analyses will be conducted with random coefficient models, a specific subset of the more general multilevel modeling framework. Statistical analyses will be conducted with the SAS computer program. The sample size supports statistical power to detect responses to intervention (i.e., effect size) of a mean change of 0.40 from baseline to follow-up.

RISKS Risks of participating in Baseline, Follow-Up, and focus group interviews are minimal. Participants could experience some discomfort providing a response to questions regarding frequency of sexual behaviors or alcohol use, or experience of HIV-related stigma, discrimination or support. Participants will be told that answering any eligibility questions or discussing topics during the focus group is entirely voluntary and that they may decide to not answer any questions at any time. Steps will be taken to ensure the anonymity of participant's self-disclosed age, sexual behaviors, and substance use for determining eligibility. All screening questions will be asked in a private setting.

There is also a risk that a bystander could overhear an IVR message or that someone else could answer the participants phone and hear an IVR message, which might result in questions to the participant about the nature or purpose of the messages. However, IVR messages are common in India, which can provide a common explanation for participants. Furthermore, participants will know when IVR calls are expected as they choose the times to receive calls and they can turn off their phones or ignore the calls if they are concerned about their privacy at any time. HIV-status disclosure will only happen if the participant chooses to disclose in response to a question from a bystander.

"National Do Not Call" registry - There are no risks to a participant who removes their cell phone number from the registry for the duration of the study.

The risk of gathering information with properly trained and supervised staff poses minimal risk to the proposed participants. Some participants may benefit from interaction with an attentive trained professional and feel good about being given a chance to express their opinions. Project staff members are trained to offer referrals to appropriate resources at the end of interviews with participants if they have heard a response that indicated that (or if they observed) the participant to be in need of services they are not otherwise receiving.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* HIV+
* Taking 1st-line ART 6 months or longer
* Missed taking any ART dose in the previous 6 months
* Able to speak and understand Bengali, Hindi, or English*
* Willing to receive health-related IVR messages on mobile phones. (If participant will use personal cell phone and is currently registered on the "National Do Not Call" (NDNC) registry, the participant must be willing to be removed from the registry for the duration of the study.)
* Able to provide informed consent
* Phase 2A - Client at MCTC or member of MNPW, or peer referral of MCTC client or MNPW member,
* Phase 2A - Received a CD4 count result in the prior two months**
* Phase 2B - Patient at Calcutta School of Tropical Medicine ART Centre, or peer referral of a patient,
* Phase 2B - Received

Exclusion Criteria:

* Less than age 18
* Not HIV+
* Not taking 1st-line ART for 6 months or longer
* Does not report missing an ART dose in the prior 6 months
* Not able to speak and understand Bengali, Hindi, or English
* Is not willing to receive health-related IVR messages on mobile phones. (If participant will use personal cell phone and is currently registered on the "National Do Not Call" (NDNC) registry, the participant is NOT willing to be removed from the registry for the duration of the study.)
* Unable to provide informed consent.
* Phase 2A - Not client at MCTC or Member of MNPW, or peer referral of MCTC client or MNPW member
* Phase 2A - Not received a CD4 count result in the prior two months
* Phase 2B - Not patient at Calcutta School of Tropical Medicine ART Centre, or peer referral of a patient,
* Phase 2B - Not received a CD4 count result in the prior month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in antiretroviral medication adherence measured by AIDS Clinical Trials Group (ACTG) self-report measure. | Change from baseline to 2-, 4-, and 6-months prospective
Change in antiretroviral medication adherence as measured by weekly IVR surveys | Change over 6 months prospective
Change in antiretroviral medication adherence as measured by pill counts at monthly medical appointments recorded in medical charts | Change from 6 months prior to baseline to 6-months prospective
Change in antiretrovial medication adherence as indicated by changes in CD4 cell counts as recorded in patients' medical charts | Change from up to 18 months before baseline to 6 months prospective

SECONDARY OUTCOMES:
Change in ART clinic appointment non-adherence resulting in lack of ART, as measured by self-report | Change from Baseline to 2-, 4-, and 6-months prospective
Change in depressive symptoms as measured by the depression subscale of the HADS self-report measure | Change from baseline to 2-, 4-, and 6-months prospective
Change in coping skills in 8 domains applied to HIV/AIDS and ART as measured by the Brief Cope self-report measure | Change from baseline to 2-, 4-, and 6-months prospective
Change in social support as measured by MOS Social Support Survey Brief 8-item self-report measure | Change from baseline to 2-, 4-, and 6-months prospective
Change in ART attitudes and adherence expectations as measured by self-report items from the ACTG measure | Change from baseline to 2-, 4-, and 6-months prospective
Change in preferences for IVR messaging as measured by self-report | 2-, 4-, and 6-months prospective
  As a pilot study, preferences and acceptability are important aims.
Change in depressive symptoms as measured 2 questions in weekly IVR surveys | Change over 6-months prospective
Change in preferences for IVR messaging as measured IVR call log data | Change over 6 months prospective
  IVR systems automatically log call information including if answered, call duration, and early termination (indicating low preference for message).
Change in preferences for IVR messaging as measured by responses to an IVR survey at the end of each IVR message | Change over 6 months prospective

OTHER OUTCOMES:
Change in physical symptoms or side effects as measured by self-report in the ACTG adherence measure. | Change from baseline to 2-, 4-, and 6-months prospective, and weekly over 6 months
  Symptom reports may indicate treatment success or failure potentially linked to adherence, and conversely, side effects may indicate medication use but also precipitate non-adherence.
Change in disclosures of HIV status as measured by self-report | Change from Baseline to 2-, 4-, and 6-months prospective
  IVR calls may result in active, passive, and inadvertent HIV+ status disclosures, which may result in improved social support or discrimination
Change in stigma related to HIV/AIDS as measured by self-report | Change from Baseline to 2-, 4-, and 6-months prospective
Change in condom Use as measured by self-report | Change from Baseline to 2-, 4-, and 6-months prospective
  Condom use is not directly targeted in the current intervention but was an original proposed study aim and may be implemented if participants request sexual health messages.
Change in alcohol consumption as measured AUDIT-C 3-item alcohol screen. | Chagne from Baseline to 2-, 4-, and 6-months prospective
  Alcohol abuse is not directly targeted in the current intervention but was an original proposed study aim and may be implemented if participants request alcohol related messages.
Change in physical symptoms or side effects as measured by one question in weekly IVR surveys. | Change over 6 months prospective
  Symptom reports may indicate treatment success or failure potentially linked to adherence, and conversely, side effects may indicate medication use but also precipitate non-adherence.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Calcutta School of Tropical Medicine ART Centre, Kokata, West Bengal
  - Durbar Mahila Samanwaya Committee (MCTC & MNPW), Kolkata, West Bengal

REFERENCES:
- [Derived] Swendeman D, Fehrenbacher AE, Roy S, Ray P, Sumstine S, Scheffler A, Das R, Jana S. A pilot randomized controlled trial (RCT) of daily versus weekly interactive voice response calls to support adherence among antiretroviral treatment patients in India. Mhealth. 2020 Oct 5;6:35. doi: 10.21037/mhealth-19-248a. eCollection 2020. PMID 33437832
- [Derived] Swendeman D, Fehrenbacher AE, Roy S, Das R, Ray P, Sumstine S, Ghose T, Jana S. Gender disparities in depression severity and coping among people living with HIV/AIDS in Kolkata, India. PLoS One. 2018 Nov 21;13(11):e0207055. doi: 10.1371/journal.pone.0207055. eCollection 2018. PMID 30462688